CLINICAL TRIAL: NCT04969874
Title: Feasibility of At Home Remote Monitoring Following a Stay in Intensive Rehabilitation in Patients with Chronic Swallowing Disorders Caused by Treatment for Cancer of the Aero-digestive Tract: Pilot Study
Brief Title: Remote Orthophonic Follow-up on Patients with Chronic Swallowing Disorders
Acronym: E-CRIL_MAX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/21/0023
Record Dates: First submitted 2021-07-08; First posted 2021-07-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Deglutition
Keywords: remote video follow-up; speech therapy; Aerodigestive cancer
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Intervention Model Description: Monocentric prospective longitudinal pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- remote follow-up (Other): patients with chronic disorders on sequelae of anti-cancer treatments after an intensive rehabilitation stay will undergo 5 months of remote follow-up with speech therapists including questionnaires and interview
  Interventions: Other: Remote follow-up

INTERVENTIONS:
Other: Remote follow-up — The feeling of swallowing will be assessed at the end of the stay at the rehabilitation center, which corresponds to the first visit, and then every month for 5 months during remote interviews and on discharge with the Deglutition Handicap Index (DHI), a self-assessment questionnaire for the swallowing handicap.
  The quality of life will be assessed at the firs visit and 6 months after using the EORTC QLQ 30 quality of life scale and the H&N annex, a self-assessment questionnaire on the quality of life for people with cancer of the head and neck.
  The satisfaction of users and the interest of city health professionals in the use of the "MAX Educ" tool as part of a monthly monitoring will be collected via the TUQ questionnaire, through the MAX platform at Month 6.

SUMMARY:
The study will assess the feasibility of monthly post rehabilitation remote monitoring, using the "MAX Educ" webvision app, in patients with sequelae of aerodigestive cancer treatments.

DETAILED DESCRIPTION:
The patients included in the study will benefit from a monthly video follow-up via the WEB tool "MAX Educ" during the first 6 months of their discharge from the rehabilitation center. They will be contacted each month during 5 months by the CRIL speech therapist for an interview (20 to 30 minutes).

The interview will take place in 2 stages; at first, a discussion phase, during which the speech therapist will take simple news of the patient. The second phase, more formal, will be the opportunity to collect the data necessary for the validation of the secondary endpoints. To do this, the speech therapist will use the Deglutition Handicap Index (DHI) and an interview grid.

The interview will be conducted using an interview sheet previously written by the project team. The following elements will be discussed: the perceived swallowing handicap (DHI), the instructions related to diet and their daily application, ongoing rehabilitation follow-ups, notable events as well as his psycho-emotional experience in relation to said disorders.

After signing the consent and verifying the eligibility criteria, all patients will be assessed upon discharge from the rehabilitation center by means of video swallowing fluoroscopy, allowing the deglutition score to be established.

EORTC Quality of Life Questionnaire (QLQ) QLQ-30 and its annex H & N35 and the DHI will also be completed at the inclusion visit at T0.

They will then be monitored monthly by video from Month 1 to Month 5.

During the end of research visit at 6 months, all the patients included will be reviewed in follow-up consultation with a doctor and a speech therapist within the intensive rehabilitation center for laryngectomees (which corresponds to the standard follow-up) and evaluated by video swallowing fluoroscopy. EORTC QLQ-30, EORTC QLQ-H & N35 quality of life questionnaires and the DHI will also have to be completed.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over and treated for cancer of the upper aero-digestive tract:
* Patient having spent a stay at the intensive rehabilitation center for laryngectomees
* Patient with a medical diagnosis of swallowing disorders at risk of inhalation
* Patient having the possibility of accessing a device allowing the use of the software by video (smartphone, tablet and / or computer)
* Informed consent signed by the patient.
* Patient affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Progressive neurological disease leading to cognitive disorders
* Patient with guardianship, curators or legal protection
* Inability to give consent
* Patient participating in another research including an exclusion period still in progress
* Patient with speech therapy whose frequency is greater than 1 weekly session

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
patient attendance at monthly remote monitoring | Month 6 : end of follow-up
  Attendance will be evaluated by measuring the rate of patients who participated in at least 3 webvisions out of 5 and at the final visit in face-to-face consultation, compared to the number of patients included.

SECONDARY OUTCOMES:
felt swallowing | Month 0 : before follow-up
  The feeling of swallowing will be evaluated with the Deglutition Handicap Index (DHI), a swallowing handicap self-assessment questionnaire. ranking from 30 to 150, 30 corresponding to no handicap swallowing, and 150 being the worst handicap to swallow
felt swallowing | Month 1 of follow-up
  The feeling of swallowing will be evaluated with the Deglutition Handicap Index (DHI), a swallowing handicap self-assessment questionnaire. ranking from 30 to 150, 30 corresponding to no handicap swallowing, and 150 being the worst handicap to swallow
felt swallowing | Month 2 of follow-up
  The feeling of swallowing will be evaluated with the Deglutition Handicap Index (DHI), a swallowing handicap self-assessment questionnaire. ranking from 30 to 150, 30 corresponding to no handicap swallowing, and 150 being the worst handicap to swallow
felt swallowing | Month 3 of follow-up
  The feeling of swallowing will be evaluated with the Deglutition Handicap Index (DHI), a swallowing handicap self-assessment questionnaire. ranking from 30 to 150, 30 corresponding to no handicap swallowing, and 150 being the worst handicap to swallow
felt swallowing | Month 4 of follow-up
  The feeling of swallowing will be evaluated with the Deglutition Handicap Index (DHI), a swallowing handicap self-assessment questionnaire. ranking from 30 to 150, 30 corresponding to no handicap swallowing, and 150 being the worst handicap to swallow
felt swallowing | Month 5 of follow-up
  The feeling of swallowing will be evaluated with the Deglutition Handicap Index (DHI), a swallowing handicap self-assessment questionnaire. ranking from 30 to 150, 30 corresponding to no handicap swallowing, and 150 being the worst handicap to swallow
felt swallowing | Month 6 of follow-up
  The feeling of swallowing will be evaluated with the Deglutition Handicap Index (DHI), a swallowing handicap self-assessment questionnaire. ranking from 30 to 150, 30 corresponding to no handicap swallowing, and 150 being the worst handicap to swallow

CONTACTS AND LOCATIONS:
Overall Officials: Anais Galtier, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No